## Title:

Clinical Evaluation of Enamel Microhardness Using At-Home and In-Office Tooth Whitening Agents

NCT#

07165366

Statistical Analysis:

April 21. 2024

## **Statistical Analysis**

Microhardness was summarized for each active treatment group and for the negative and positive controls. Microhardness comparisons for the treatments and negative controls were performed using ANOVA, with a fixed effect for treatment and a random effect to account for within-subject correlations. Pair-wise tests between treatments were performed using the Sidak method to control the overall significance level. Shade change was summarized by treatment and compared between treatments using Wilcoxon Signed Rank tests (at-home versus in-office) and Wilcoxon Rank Sum tests (at-home with versus without PF). A two-sided overall 5% significance level was used.